CLINICAL TRIAL: NCT04992533
Title: Tourniquet vs. no Tourniquet During High Tibial Osteotomy：A Randomized Controlled Trial
Brief Title: Tourniquet vs. no Tourniquet During High Tibial Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Qilu200326
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-duration tourniquet (Active Comparator): Tourniquets inflated before arthroscopic exploration and deflated after high tibial osteotomy
  Interventions: Procedure: Long-duration tourniquet
- Short-duration tourniquet (Experimental): Tourniquet should be inflated before arthroscopic exploration and deflated immediately after the exploration
  Interventions: Procedure: Short-duration tourniquet

INTERVENTIONS:
Procedure: Long-duration tourniquet — Tourniquet is used in arthroscopic exploration and high tibial osteotomy
  Arms: Long-duration tourniquet
Procedure: Short-duration tourniquet — Tourniquet is only used for arthroscopic exploration
  Arms: Short-duration tourniquet

SUMMARY:
The purpose of this study is to correlate functional outcomes and perioperative complications with tourniquet use during high tibial osteotomy.

DETAILED DESCRIPTION:
Tourniquet is widely used in orthopedic surgery, but its effect and safety in high tibial osteotomy have not been studied. This study evaluated the efficacy and safety of tourniquets by comparing different timing of use.Investigators aimed to quantify the effect of tourniquet use on reducing blood loss and to evaluate the impact of tourniquet use on functional and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* 1.Simple knee medial compartment osteoarthritis High tibial osteotomy.
* 2. With varus deformity, medial proximal tibia angle <85°
* 3. Unilateral High tibial osteotomy
* 4. Informed consent: Participants must be able to understand and voluntarily sign a written informed consent and follow the research protocol and interview process

Exclusion Criteria:

* 1.Patients who underwent other knee surgery within 6 months
* 2.Preoperative combined anemia (Hb<100g/l)
* 3.Patients with severe cardiovascular, hepatic, renal and hematopoietic diseases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | within operation
  The calculation of intraoperative blood loss includes the fluid in the aspirator bottle minus the flushing fluid used in the operation, plus the net weight added by the gauze pad weighing
Postoperative blood loss | The third day after operation
  Total blood loss preoperative blood volume =(preoperative hematocrit-postoperative Hematocrit) + transfusion volume.
Volume of drainage | Postoperative Day One
  Reactive blood loss
Thigh pain measured by Visual Analogue Scale Postoperative Day 1 | 1 day after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Thigh pain measured by Visual Analogue Scale Postoperative Day 2 | 2 day after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Thigh pain measured by Visual Analogue Scale Postoperative Day 3 | 3 day after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Thigh pain measured by Visual Analogue Scale Postoperative Day 5 | 5 day after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Thigh pain measured by Visual Analogue Scale Postoperative Week 1 | 1 week after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Thigh pain measured by Visual Analogue Scale Postoperative Week 4 | 4 week after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Thigh pain measured by Visual Analogue Scale Postoperative Week 12 | 12 week after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Crus pain measured by Visual Analogue Scale Postoperative Day 1 | 1 day after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Crus pain measured by Visual Analogue Scale Postoperative Day 2 | 2 day after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Crus pain measured by Visual Analogue Scale Postoperative Day 3 | 3 day after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Crus pain measured by Visual Analogue Scale Postoperative Day 5 | 5 day after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Crus pain measured by Visual Analogue Scale Postoperative Week 1 | 1 week after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Crus pain measured by Visual Analogue Scale Postoperative Week 4 | 4 week after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.
Crus pain measured by Visual Analogue Scale Postoperative Week 12 | 12 week after surgery
  Draw a 10 cm horizontal line on the paper. One end of the line is 0, indicating no pain; the other end is 10, indicating severe pain; and the middle part indicates varying degrees of pain. The patient selects a point from the horizontal line and the length from 0 to this point is the Visual Analogue Scale score.

CONTACTS AND LOCATIONS:
Overall Officials: Peilai Liu, MD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
The datasets used and/or analysed during the current study are available from the overall study officials on reasonable request.

REFERENCES:
- [Background] Goel R, Rondon AJ, Sydnor K, Blevins K, O'Malley M, Purtill JJ, Austin MS. Tourniquet Use Does Not Affect Functional Outcomes or Pain After Total Knee Arthroplasty: A Prospective, Double-Blinded, Randomized Controlled Trial. J Bone Joint Surg Am. 2019 Oct 16;101(20):1821-1828. doi: 10.2106/JBJS.19.00146. PMID 31626006
- [Background] Jawhar A, Stetzelberger V, Kollowa K, Obertacke U. Tourniquet application does not affect the periprosthetic bone cement penetration in total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2019 Jul;27(7):2071-2081. doi: 10.1007/s00167-018-5330-7. Epub 2018 Dec 11. PMID 30539303
- [Background] Wang K, Ni S, Li Z, Zhong Q, Li R, Li H, Ke Y, Lin J. The effects of tourniquet use in total knee arthroplasty: a randomized, controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Sep;25(9):2849-2857. doi: 10.1007/s00167-015-3964-2. Epub 2016 Jan 8. PMID 26745962